CLINICAL TRIAL: NCT05063591
Title: Removing Transfusion Dependence as a Barrier to Hospice Enrollment
Acronym: BRUOG-407
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adam Olszewski (Other)
Responsible Party: Sponsor-Investigator, Adam Olszewski, Associate Professor of Medicine, Brown University
Organization: Brown University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BRUOG-407
Record Dates: First submitted 2021-09-11; First posted 2021-10-01 (Actual); Results first posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Hematologic Malignancy; Myelodysplastic Syndromes; Acute Myeloid Leukemia; Lymphoma; Leukemia; Myeloma
Keywords: palliative care
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Lymphoma; Leukemia; Neoplasms, Plasma Cell

STUDY DESIGN:
Intervention Model Description: single-center, prospective pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Patients with aggressive hematologic malignancies who are hospice eligible, not pursuing further cancer directed therapy, and whose primary hematologist is planning to initiate a conversation regarding transition to hospice will be eligible for enrollment.
  Interventions: Other: Transfusion support

INTERVENTIONS:
Other: Transfusion support — Patients will be offered symptom-driven transfusion support in addition to standard hospice care

SUMMARY:
Hospice care at the end of life (EOL) includes a multidisciplinary team that helps patients and families focus on symptom control and quality of life. For patients with "solid" (e.g. lung, breast) cancers it has been shown to improve quality of life for both patients and families. Unfortunately, patients with blood cancers (e.g. leukemia, lymphoma) often delay their enrollment and receive more aggressive care at the EOL. One factor in this delay is the inability for patients to receive blood transfusions while on hospice. Patients with blood cancers often require frequent blood transfusions near the EOL for symptom control. The structure of Medicare hospice benefit makes coverage for transfusions financially unfeasible for hospice agencies, and therefore patients with blood cancers will delay enrollment onto hospice in order to continue to receive blood transfusions.

The objective of this study is to evaluate whether removing this financial burden, through external funding of blood transfusions for patients while on hospice, will encourage patients with blood cancers to enroll on hospice earlier and ultimately improve their and their caregivers EOL care.

DETAILED DESCRIPTION:
The overall objective is to demonstrate the feasibility of providing blood transfusions to patients with HM enrolled on hospice, and to evaluate both EOL care quality outcomes in these patients, and caregiver quality of life and perception of patient EOL care quality. Palliative blood transfusions will be provided to patients on this study free of cost through study funding. The hypothesis is that removing transfusion dependence as a barrier to hospice enrollment for patients with hematologic malignancies will result in improved EOL care quality outcomes. This hypothesis is derived from our previous research demonstrating that for Medicare beneficiaries with HM, transfusion dependence poses a significant barrier to timely hospice referral.

The study design is to conduct a single-center, prospective pilot study . Patients with aggressive hematologic malignancies who are hospice eligible, not pursuing further cancer directed therapy, and whose primary hematologist is planning to initiate a conversation regarding transition to hospice will be pursued for enrollment. These patients will be offered to enroll in this study in which funding will be provided to receive palliative blood transfusions while enrolled on hospice.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and older
* Advanced hematologic malignancies
* Hospice eligible as determined by their primary hematologist
* Have opted to forego further cancer-directed therapy.
* Transfusion Dependent: Requiring at least 2 units of blood products

Exclusion Criteria:

* Patients with major psychiatric illness
* Patients without the ability to speak and read English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-07-09 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela C Egan, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Cancer Research and Clinical Trials at Lifespan Cancer Institute — https://www.lifespan.org/centers-services/cancer-research-and-clinical-trials

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 22 patients and 9 caregivers screened, 10 patients (45%) and 8 caregivers enrolled. 4 screened patients died before consenting.
Groups:
- Caregivers: Patient caregivers
Period: Overall Study
Arm/Group | Intervention Arm | Caregivers
Started | 10 | 8
Completed | 10 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Caregivers: Caregivers of participants in Arm A
- Total: Total of all reporting groups
Arm/Group | Intervention Arm | Caregivers | Total
Number analyzed (Participants) | 10 | 8 | 18
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 80 [77 to 84] | 60 [55 to 77] | 77.5 [62 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 6 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Diagnosis [Count of Participants; unit: Participants] — Only relevant to the Intervention Arm Population: Caregivers do not have a diagnosis, so 0 participants from that arm have been analyzed and they are not included in the total
  Participants
    number analyzed (Participants) | 10 | 0 | 10
    Acute myeloid leukemia | 6 | 0 | 6
    Other | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eligible Patients Choosing to Participate in the Care Model Under Study Rather Than Standard of Care.
Description: Measured as: the number of eligible patients approached and number who elect to enter the study and participate in the novel care model rather than through the traditional hospice care model.
Time Frame: Through study completion, on average 2 years
Population: Eligible patients approached for participation
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 22
Participants | 10

2. Secondary Outcome: Time Enrolled on Hospice.
Description: Count endpoint: number of days enrolled on hospice
Time Frame: From enrollment until death or withdrawal of consent, on average 2 months.
Measure: Median (Full Range); unit: days
Arm/Group | Intervention Arm
Number analyzed (Participants) | 10
days | 13 [4 to 103]

3. Secondary Outcome: Number of Days in the ICU in the Last 30 Days of Life
Description: Count endpoint: Number of days subject spent in the ICU in the last 30 days of life
Time Frame: Last 30 days of life.
Measure: Median (Full Range); unit: days
Arm/Group | Intervention Arm
Number analyzed (Participants) | 10
days | 0 [0 to 0]

4. Secondary Outcome: Death in an Acute Care Hospital
Description: Binary endpoint: met if subject passed away in an acute care hospital
Time Frame: From enrollment until death or withdrawal of consent, on average 2 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 10
Participants | 0

5. Secondary Outcome: Receipt of Chemotherapy in the Last 14 Days of Life
Description: Binary endpoint: met if subject received chemotherapy in the last 14 days of life
Time Frame: Last 14 days of life
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: From the date of study enrollment until the date of death.
Description: Information about adverse effects associated with blood transfusions were collected, only for participants in Arm A (Intervention Arm). Adverse events in the "Caregiver" arm were not collected.
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 10/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT05063591/Prot_SAP_000.pdf